CLINICAL TRIAL: NCT05468476
Title: Multi-omics Analysis of Women With PCOS and Obesity Compared With Non-PCOS Obese Controls
Status: Completed | Type: Observational
Sponsor: Zhang Manna (Other)
Responsible Party: Sponsor-Investigator, Zhang Manna, Director, Principal Investigator, Clinical Professor, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: Multi-omics PCOS
Record Dates: First submitted 2022-05-18; First posted 2022-07-21 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Gut microbiome; metabolomics; transcriptomic; obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Metabolome Serum Sample Collection，Transcriptome RNA sample collection and Stool specimen collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with PCOS (PCOS group): PCOS women with obesity previously diagnosed with PCOS（meet the 2003 Rotterdam diagnostic criteria） not using hormonal therapy and without other significant health or endocrine issues.
  Interventions: Other: No intervention
- Women without PCOS (Non-PCOS group): This study enrolled age- and body mass index (BMI)-matched subjects with normal menstrual cycles, not using hormonal therapy, and without any significant health or endocrine issues.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine and metabolic disorder in reproductive-aged women， which associated with increased risks to develop metabolic disorders, including cardiovascular diseases, diabetes mellitus, and cerebrovascular diseases. The precise pathogenesis of PCOS remains unknown but is thought to be multifactorial, comprising genetic and environmental factors .

DETAILED DESCRIPTION:
To study the pathogenesis of diseases, the study of multi-omics approach has been applied in various diseases researching . Obesity and PCOS are both metabolic disorders, and both have an impact on metagenomics, metabolomics and transcriptome. Currently, multi-omics studies based on obese PCOS are still limited. Therefore, this study tried to use a multi-omics approach that integrates the gut microbiome, serum metabolomics, serum transcriptomics, and clinical indicators to distinguish obese PCOS from obese non-PCOS women. To investigate whether the specific composition of the gut microbiome is associated with PCOS in obese women. Serum metabolomics and transcriptomics were analyzed to explore potential metabolic pathways. Meanwhile, gut microbiome and serum metabolomics are used to predict the occurrence of PCOS. Then, a new metabolite that could predict PCOS were tested on female mice with high fat diet (HFD).

ELIGIBILITY:
Inclusion Criteria:

* patients with obesity (BMI>28kg/m2)
* aged 18-45 years
* Diagnosis of PCOS
* the Rotterdam diagnosis criteria (2003)

Exclusion Criteria:

* Pregnant women;
* Hyperthyroidism or hypothyroidism
* Severe liver and kidney function injury
* Cancer patients;
* Associated with severe infection, severe anemia, neutropenia and other blood system diseases;
* Have type 1 diabetes, single-gene mutated diabetes or other secondary diabetes;
* Patients with mental illness or intellectual disability;
* Have taken drugs for PCOS treatment in the last three months;
* Taking drugs or foods (antibiotics, probiotics, yogurt, etc.) that affect the intestinal flora for nearly one month;
* Have a long history of taking hormone therapy;
* Currently or recently participating in another clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study enrolled 63 PCOS women with obesity and 58 age- and body mass index (BMI)-matched subjects with normal menstrual cycles who were admitted to the Department of Endocrinology, Shanghai Tenth People's Hospital, between April 2019 and November 2022.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Phenotype differences in the Serum non-targeted metabolomics by LC-MS. | Samples to be collected once per participant within 7 days of enrollment.
  Understand phenotypical differences from biological samples comparing women with and without PCOS. Venipuncture blood draws are to be completed and analyzed by a commercial laboratory to comprehensively analyze non-target metabolites.
Phenotype differences in the gut microbiome by metagenomic sequencing. | Samples to be collected once per participant within 7 days of enrollment
  Understand phenotypical differences from biological samples comparing women with and without PCOS. Stool samples are to be collected by women and analyzed with metagenomics sequencing.
Phenotype differences in the transcriptome expression by mRNA-seq. | Samples to be collected once per participant within 7 days of enrollment.
  Understand phenotypical differences from biological samples comparing women with and without PCOS. The researcher will collect and analyze Venipuncture blood for RNA. Differences in the expression of genes between the two groups of subjects, analysis to select possible pathogenic factors leading to the pathogenesis of PCOS.
Phenotype differences in the Serum targeted metabolomics by LC-MS. | Samples to be collected once per participant within 7 days of enrollment.
  Understand phenotypical differences from biological samples comparing women with and without PCOS. Venipuncture blood draws are to be completed and analyzed by a commercial laboratory to comprehensively analyze the target metabolite.

SECONDARY OUTCOMES:
BMI | Samples to be collected once per participant within 7 days of enrollment.
  Body mass index (BMI)=weight(kg)/height(m)^2.
TT | Samples to be collected once per participant within 7 days of enrollment.
  total testosterone in nmol/L.
LH | Samples to be collected once per participant within 7 days of enrollment.
  luteinizing hormone in IU/L.
FSH | Samples to be collected once per participant within 7 days of enrollment.
  The follicle-stimulating hormone in IU/l.
E2 | Samples to be collected once per participant within 7 days of enrollment.
  Estradiol in pmol/L.
PRL | Samples to be collected once per participant within 7 days of enrollment.
  Prolactin in uIU/ml.
HC | Samples to be collected once per participant within 7 days of enrollment.
  Hip Circumference in centimeters.
WC | Samples to be collected once per participant within 7 days of enrollment.
  Waist Circumference in centimeters.
Waist/hip Ratio | Samples to be collected once per participant within 7 days of enrollment.
  WHR=(Waist Circumference in centimeters)/(Hip Circumference in centimeters).
Menstrual cycles | Samples to be collected once per participant within 7 days of enrollment.
  the total number of menstrual periods in the last year.
FBG | Samples to be collected once per participant within 7 days of enrollment.
  fasting blood-glucose in mmol/L.
PBG | Samples to be collected once per participant within 7 days of enrollment.
  postprandial blood-glucose in mmol/L.
FINS | Samples to be collected once per participant within 7 days of enrollment.
  fasting serum insulin in mU/L.
PINS | Samples to be collected once per participant within 7 days of enrollment.
  postprandial insulin in mU/L.
ALT | Samples to be collected once per participant within 7 days of enrollment.
  alanine aminotransferase in U/L.
AST | Samples to be collected once per participant within 7 days of enrollment.
  aspartate aminotransferase in U/L.
UA | Samples to be collected once per participant within 7 days of enrollment.
  Uric acid in umol/L.
CR | Samples to be collected once per participant within 7 days of enrollment.
  Creatinine in umol/L.
Ferriman-Gallwey score | Samples to be collected once per participant within 7 days of enrollment.
  The minimum value of Ferriman-Gallwey score is 0 and the maximum value is 44. An Ferriman-Gallwey score greater than or equal to 6 is considered to be a clinical manifestation of androgen excess.
HOMA-IR | Samples to be collected once per participant within 7 days of enrollment.
  Homeostatic model assessment insulin resistance index=FBG*FINS/22.5.
HbA1c (%) | Samples to be collected once per participant within 7 days of enrollment.
  glycosylated hemoglobin (%).
γ-GT | Samples to be collected once per participant within 7 days of enrollment.
  γ-glutamyl transferase in U/L.
BUN | Samples to be collected once per participant within 7 days of enrollment.
  urea nitrogen in mmol/L.
SOD | Samples to be collected once per participant within 7 days of enrollment.
  Superoxide dismutase in pg/ml.
Interleukin 22, IL-22 | Samples to be collected once per participant within 7 days of enrollment.
  Interleukin 22 in pg/ml. The factor reflects that the organism is in an inflammatory state. There is no maximum or minimum value for the factor and the higher scores mean a worse outcome.
Interleukin 6，IL-6 | Blood samples to be collected once per participant within 7 days of enrollment.
  Interleukin 6 in pg/ml. The factor reflects that the organism is in an inflammatory state. There is no maximum or minimum value for the factor and the higher scores mean a worse outcome.
Interleukin 8， IL-8 | Blood samples to be collected once per participant within 7 days of enrollment.
  Interleukin 8 in pg/ml. The factor reflects that the organism is in an inflammatory state. There is no maximum or minimum value for the factor and the higher scores mean a worse outcome.
Tumor Necrosis Factor， TNF | Blood samples to be collected once per participant within 7 days of enrollment.
  Tumor Necrosis Factor in pg/ml. The factor reflects that the organism is in an inflammatory state. There is no maximum or minimum value for the factor and the higher scores mean a worse outcome.
FT | Blood samples to be collected once per participant within 7 days of enrollment.
  free testosterone in nmol/L.
DHEAS | Blood samples to be collected once per participant within 7 days of enrollment.
  Dehydroepiandrosterone Sulfate in ug/dl.
SHBG | Blood samples to be collected once per participant within 7 days of enrollment.
  sex hormone-binding globulin in nmol/L.
AD | Blood samples to be collected once per participant within 7 days of enrollment.
  Androstenedione in ng/ml.
LDL-c | Blood samples to be collected once per participant within 7 days of enrollment.
  low-density lipoprotein cholesterol in mmol/L.
HDL-c | Blood samples to be collected once per participant within 7 days of enrollment.
  high-density lipoprotein cholesterol in mmol/L.
TC | Blood samples to be collected once per participant within 7 days of enrollment.
  Total Cholesterol in mmol/L.
TG | Blood samples to be collected once per participant within 7 days of enrollment.
  Triglyceride in mmol/L.
CRP | Blood samples to be collected once per participant within 7 days of enrollment.
  C reactive protein in pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Manna Zhang, Ph.D, Principal Investigator — Department of Endocrinology, Shanghai Tenth People's Hospital
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No